CLINICAL TRIAL: NCT01473407
Title: A Therapeutic-equivalence Study Comparing The Efficacy And Safety Of Intravenous Epoetin Hospira And Epoetin Alfa (Amgen) In Patients With Chronic Renal Failure Requiring Hemodialysis And Receiving Epoetin Maintenance Treatment
Brief Title: A Phase 3 Study Comparing the Effects of Intravenous Epoetin Hospira and Epoetin Alfa [Epogen] (Amgen) in Patients With Chronic Renal Failure Requiring Hemodialysis and Receiving Epoetin Maintenance Treatment. AiME - Anemia Management With Epoetin
Acronym: AiME - 01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPOE-10-01; C3461001 (Other: Alias Study Number)
Record Dates: First submitted 2011-11-02; First posted 2011-11-17 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Chronic Kidney Disease; Chronic Renal Failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epoetin Hospira (Experimental): Epoetin Hospira
  Interventions: Biological: Epoetin Hospira
- Epogen (Amgen) (Active Comparator): Epogen (Amgen)
  Interventions: Biological: Epogen (Amgen)

INTERVENTIONS:
Biological: Epoetin Hospira — Variable dose
  Arms: Epoetin Hospira
Biological: Epogen (Amgen) — Variable dose
  Other Names: Epoetin Alfa
  Arms: Epogen (Amgen)

SUMMARY:
The purpose of this study is to demonstrate therapeutic equivalence of IV Epoetin Hospira compared to IV Epogen (Amgen), based on maintenance of Hb levels and study drug dose requirements in patients treated for anemia associated with chronic renal failure and on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to provide written informed consent after risks and benefits of the study have been explained prior to any study related activities
2. Hemodialysis patients with chronic renal failure and renal anemia currently on stable Epogen (Amgen) treatment for at least 4 weeks prior to randomization, for whom the following apply (during this period):

   * Epogen (Amgen) dose has been administered intravenously 1 to 3 times per week with no more than a 10% dose change from the mean for at least 4 weeks prior to randomization
   * Stable hemoglobin, defined as meeting all of the following:

     * Mean hemoglobin during the 4 weeks prior to randomization between 9.0 and 11.0 g/dL
     * No more than one hemoglobin outside of range from 9.0-11.0 g/dL during the 4 weeks prior to randomization
     * No hemoglobin result more than ±1 g/dL from the mean hemoglobin level during the 4 week period prior to randomization
3. Patients on stable, adequate dialysis for at least 12 weeks prior to randomization, defined as no clinically relevant changes of dialysis regimen and/or dialyzer
4. Patients with adequate iron stores, defined as ferritin >100 μg/L and TSAT >20%, prior to randomization
5. Male or female patients aged 18 to 80 years (both inclusive)
6. If female, patient must be either postmenopausal for at least 1 year prior to randomization, surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or practicing at least 1 of the following methods of birth control:

   * hormonal contraceptives (oral, parenteral, or transdermal) for at least 3 months prior to randomization
   * intrauterine device (IUD)
   * double-barrier method (condoms, contraceptive sponge, diaphragm, or vaginal ring with spermicidal jellies or cream)

If hormonal contraceptives are used, the specific contraceptive must have been used for at least 3 months prior to randomization. If the patient is currently using a hormonal contraceptive, she should also use a barrier method during this study and for at least 30 days following the administration of the patient's last dose

Exclusion Criteria:

1. Maintenance Epoetin dosage >600 U/kg per week (1-3 times per week)
2. Treatment with long-acting epoetin analogues such as Aranesp ® within 3 months prior to randomization
3. Any of the following within 3 months prior to randomization:

   * Myocardial infarction
   * Stroke (cerebrovascular accident)/cerebrovascular insult (minor stroke) or transient ischemic attack/intracerebral bleeding/cerebral infarction
   * Severe/unstable angina
   * Coronary angioplasty, bypass surgery, or peripheral artery bypass graft
   * Decompensated congestive heart failure (New York Heart Association [NYHA] class IV)
   * Pulmonary embolism
   * Deep vein thrombosis or other thromboembolic event
   * Received live or attenuated vaccination (except flu vaccination)
4. Uncontrolled Hypertension within the 4 weeks prior to randomization, defined as more than 10% of post-dialysis blood pressures >170 mmHg systolic and/or >110 mmHg diastolic, based on blood pressure readings obtained when the patient's post-dialysis body weight was not more than 0.5 kg above their listed dry weight
5. Known, clinically manifested deficiency of folic acid and/or vitamin B12 (irrespective of whether currently treated or not)
6. A patient with any active, uncontrolled systemic, inflammatory or malignant disease (including demyelinating diseases such as multiple sclerosis) that in the Investigator's opinion may be significant to exclude participation in the study, including but not limited to microbial, viral, or fungal infection or mental disease
7. Contraindication for the test drug or have been previously treated with Epoetin Hospira
8. Relative or absolute iron deficiency prior to randomization
9. Platelet count below 100 x 10^9/L
10. Clinically relevant increase of CRP (>10 mg/dL) for at least 2 weeks
11. Significant drug sensitivity or a significant allergic reaction to any drug, as well as known hypersensitivity or idiosyncratic reaction to epoetin (or its excipients, including albumin) or any other related drugs that in the judgment of the Investigator is exclusionary for the study participation
12. History of any of the following:

    * Detectable anti- rhEPO antibodies
    * Clinically relevant malnutrition
    * Confirmed aluminum intoxication
    * Myelodysplastic syndrome
    * Known bone marrow fibrosis (osteitis fibrosa cystica)
    * Known seizure disorder
    * Liver cirrhosis with clinical evidence of complications (portal hypertension, splenomegaly, ascites)
13. A female patient who is pregnant, lactating or planning a pregnancy during the study
14. History of drug abuse or alcohol abuse within 2 years prior to randomization as determined by the Investigator
15. Current participation or participation in a drug or other investigational research study within 30 days prior to randomization
16. May not be able to comply with the requirements of this clinical study, communicate effectively with study personnel, or is considered by the Investigator, for any reason, to be an unsuitable candidate for the study
17. Donated or lost >475 mL (i.e., 1 pint) blood volume (including plasmapheresis) or had a transfusion of any blood product within 3 months prior to randomization
18. A patient who in the Investigator's opinion, has any clinically significant abnormal laboratory evaluations, including liver function taken at Screening Visit
19. Positive laboratory test for human immunodeficiency virus (HIV) or hepatitis B surface antigen (HBsAg)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2012-01-31 (Actual); Primary Completion 2014-02-11 (Actual); Study Completion 2014-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (85):
- United States (84):
  - Montgomery Kidney Specialists, Montgomery, Alabama
  - Southwest Clinical Research Institute, LLC, Tempe, Arizona
  - Lakhi M. Sakhrani, MD A Medical Coporation, Alhambra, California
  - North America Research Institute, Azusa, California
  - DaVita Dialysis Center-Bakersfield Dialysis Center, Bakersfield, California
  - Ong, Rubin, Shahmir A Medical Corp DBA: Solano Kidney Care, Fairfield, California
  - A Medical Corporation, Glendale, California
  - Renal Consultants Medical Group, Granada Hills, California
  - La Puente Dialysis Center, La Puente, California
  - Advanced Medical Research, LLC, Lakewood, California
  - DaVita Bixby Knolls Dialysis, Long Beach, California
  - Bayview Nephrology, Inc, Long Beach, California
  - Academic Medical Research Institute, Los Angeles, California
  - Desert Nephrology Medical Group, Modesto, California
  - La Jolla Clinical Research, Inc., National City, California
  - Valley Renal Medical Group, Northridge, California
  - Ontario Dialysis Inc, Ontario, California
  - Discovery medical Research Group, Inc., Porterville, California
  - Nephrology Educational Services and Research, Inc, Tarzana, California
  - Queen Dialysis Center, West Covina, California
  - American Institute of Research, Whittier, California
  - Mark C. Lee, Inc. Santa Fe Springs Dialysis, Whittier, California
  - North Valley Nephrology, Yuba City, California
  - Nephrology and Hypertension Associates, Middlebury, Connecticut
  - South Florida Nephrology, Inc., Coral Springs, Florida
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - San Marcus Research Clinic, Inc, Miami, Florida
  - Nephrology Associates of South Miami, Miami, Florida
  - ARA Naples South Dialysis Center, Naples, Florida
  - ARA- Naples Dialysis Center, LLC, Naples, Florida
  - Innovative Medical Research of South Florida, Inc., North Miami Beah, Florida
  - Discovery Medical Research Group, Inc., Ocala, Florida
  - Central Florida Kidney Centers, Orlando, Florida
  - Renal Physicians of Georgia, PC, Dublin, Georgia
  - Boise Kidney & Hypertension Institute, PLLC, Meridian, Idaho
  - Research by Design, LLC, Evergreen Park, Illinois
  - North Suburban Nephrology, LLC, Gurnee, Illinois
  - Nephrology Specialists, PC, Merrillville, Indiana
  - Westbank Nephrology Associates, Marrero, Louisiana
  - Internal Medicine Specialists, New Orleans, Louisiana
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - DaVita Dialysis Centers, Clinton Township, Michigan
  - St. Clair Specialty Physicians, P.C., Detroit, Michigan
  - South Mississippi Medical Research, PLLC, Gulfport, Mississippi
  - Chromalloy American Kidney Center, St Louis, Missouri
  - Kidney Specialists of Southern Nevada, Las Vegas, Nevada
  - Hypertension & Nephrology Associates, Eatontown, New Jersey
  - Brookdale Physician Dialysis Associates, Brooklyn, New York
  - Lower Manhattan Dialysis Center, New York, New York
  - Mountain Kidney and Hypertension Associates, PA, Asheville, North Carolina
  - East Carolina University, ECU School of Medicine, Department of Internal Medicine, Greenville, North Carolina
  - Eastern Nephrology Associates, PLLC, New Bern, North Carolina
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - HNC Dialysis Ltd., Columbus, Ohio
  - Bayview Nephrology, Inc, Erie, Pennsylvania
  - DaVita-Erie Dialysis Center, Erie, Pennsylvania
  - UPMC Hamot Clinical Trials Department, Erie, Pennsylvania
  - Franklin Dialysis Center, Philadelphia, Pennsylvania
  - Delaware Valley Nephrology and Hypertension Associates, PC, Philadelphia, Pennsylvania
  - Nephrology and Internal Medicine of Anderson, Anderson, South Carolina
  - Columbia Nephrology Associates, P.A., Columbia, South Carolina
  - Columbia Nephrology Associates, PA, Columbia, South Carolina
  - Palmetto Nephrology, PA, Orangeburg, South Carolina
  - South Carolina Nephrology and Hypertension Center, Inc., Orangeburg, South Carolina
  - Desert Nephrology Medical Group, Sumter, South Carolina
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - South Arlington Dialysis Center, Arlington, Texas
  - Texas Renal Care, Greenville, Texas
  - Med Center Dialysis, Houston, Texas
  - Meyerland Dialysis, Houston, Texas
  - Millenium Clinical Research, Inc., Houston, Texas
  - Millennium Clinical Research, Inc., Houston, Texas
  - Research Across America, Houston, Texas
  - Southwest Houston Dialysis, Houston, Texas
  - Southwest Houston Research, Ltd., Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Private practice of Roberto Mangoo-Karim MD, McAllen, Texas
  - Missouri City Dialysis, Missouri City, Texas
  - San Antonio Kidney Disease Center Physicians Group, P.L.L.C., San Antonio, Texas
  - DaVita Dialysis Center-Floyd Curl Dialysis, San Antonio, Texas
  - Clinical Research and Consulting Center, LLC, Fairfax, Virginia
  - Peninsula Kidney Associates, Hampton, Virginia
  - Internal Medicine Kidney and Hypertension Center, Norfolk, Virginia
- Consolidated Medical Plaza, Caguas, Puerto Rico

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Wish JB, Rocha MG, Martin NE, Reyes CRD, Fishbane S, Smith MT, Nassar G. Long-term Safety of Epoetin Alfa-epbx for the Treatment of Anemia in ESKD: Pooled Analyses of Randomized and Open-label Studies. Kidney Med. 2019 Aug 28;1(5):271-280. doi: 10.1016/j.xkme.2019.06.009. eCollection 2019 Sep-Oct. PMID 32734207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with chronic renal failure were receiving Epoetin maintenance therapy prior to enrollment and treatment in this study.
Groups:
- Epoetin Hospira: Participants were enrolled to receive intravenous (IV) injection of Epoetin Hospira 1 to 3 times every week over a period of 24 weeks. Dose was adjusted to maintain the hemoglobin (Hb) level from 9 to 11 gram per deciliter (g/dL). Participants were followed up to Week 28.
- Epogen: Participants were enrolled to receive IV injection of Epogen 1 to 3 times every week over a period of 24 weeks. Dose was adjusted to maintain the Hb level from 9 to 11 g/dL. Participants were followed up to Week 28.
Period: Overall Study
Arm/Group | Epoetin Hospira | Epogen
Started | 306 | 306
Completed | 252 | 259
Not Completed | 54 | 47
Not completed — Physician Decision | 1 | 4
Not completed — Lost to Follow-up | 10 | 4
Not completed — Adverse Event | 8 | 8
Not completed — Randomization Error | 3 | 1
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Kidney Transplant | 7 | 6
Not completed — Vacation/Travel | 1 | 1
Not completed — Elevated Hemoglobin | 1 | 0
Not completed — Patient Received Aranesp | 1 | 0
Not completed — Patient Lost Green Card Status | 1 | 0
Not completed — Temperature Excursion | 2 | 3
Not completed — Transfer to Another Facility/Unit | 4 | 3
Not completed — Sponsor's Decision | 10 | 10
Not completed — Site Closure | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Epoetin Hospira | Epogen | Total
Number analyzed (Participants) | 306 | 306 | 612
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.32 (13.057) | 57.35 (11.440) | 56.34 (12.307)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 131 | 277
  Male | 160 | 175 | 335

OUTCOME MEASURES:

1. Primary Outcome: Mean Weekly Hemoglobin Level From Week 21 to Week 24
Time Frame: Week 21 up to Week 24
Population: ITT population included all participants who were randomized to study treatment.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 306 | 306
g/dL | 10.17 (0.847) | 10.28 (0.839)
Statistical Analysis 1: Comparison: Epoetin Hospira vs Epogen; Least Square (LS) mean and 95 percent confidence interval (CI) were derived from an ANCOVA model with fixed effect of treatment; Test type: Non-Inferiority or Equivalence — An equivalence margin of +/- 0.5 was considered relevant to demonstrate the equivalence of the two products; LS Mean Difference = -0.12, 95% CI 2-sided [-0.25 to 0.01], Standard Error of Mean 0.066

2. Primary Outcome: Mean Weekly Dosage of Study Medication From Week 21 to Week 24
Time Frame: Week 21 up to Week 24
Population: ITT population included all participants who were randomized to study treatment. Here, "Number of Participants Analyzed (N)" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: unit per kilogram per week (U/kg/week)
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 305 | 305
unit per kilogram per week (U/kg/week) | 89.61 (99.824) | 90.37 (88.492)
Statistical Analysis 1: Comparison: Epoetin Hospira vs Epogen; LS mean and 95 percent CI were derived from an ANCOVA model with fixed effect of treatment; Test type: Non-Inferiority or Equivalence — An equivalence margin of +/- 0.5 was considered relevant to demonstrate the equivalence of the two products; LS Mean Difference = 0.37, 95% CI 2-sided [-10.40 to 11.13], Standard Error of Mean 5.483

3. Secondary Outcome: Mean Weekly Hemoglobin Level Through 24 Weeks
Time Frame: Week 1 up to Week 24
Population: ITT population included all participants who were randomized to study treatment. Here, "N" signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 302 | 305
g/dL | 10.25 (0.591) | 10.26 (0.597)
Statistical Analysis 1: Comparison: Epoetin Hospira vs Epogen; Test type: Superiority or Other; p = 0.7563, Wilcoxon Rank Sum test — P-value was calculated from a Wilcoxon Rank Sum test and t-approximation was used

4. Secondary Outcome: Mean Weekly Dosage of Study Medication Through 24 Weeks
Time Frame: Week 1 up to Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/kg/week
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 301 | 305
U/kg/week | 87.51 (86.405) | 90.95 (80.619)
Statistical Analysis 1: Comparison: Epoetin Hospira vs Epogen; Test type: Superiority or Other; p = 0.1061, Wilcoxon Rank Sum test — P-value was calculated from a Wilcoxon Rank Sum test and t-approximation was used

5. Secondary Outcome: Total Dose of Study Medication Administered
Time Frame: Week 1 up to Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units of study medication
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 301 | 305
units of study medication | 146752.6 (156128.97) | 147145.2 (141911.73)
Statistical Analysis 1: Comparison: Epoetin Hospira vs Epogen; Test type: Superiority or Other; p = 0.3369, Wilcoxon Rank Sum test — P-value was calculated from a Wilcoxon Rank Sum test and t-approximation was used

6. Secondary Outcome: Percentage of Participants With Mean Weekly Hemoglobin Level Within the Target Range
Description: Percentage of participants who had hemoglobin level within the target range of 9 to 11 g/dL for the specified weeks were reported.
Time Frame: Week 12, 24
Population: ITT population included all participants who were randomized to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 306 | 306
percentage of participants
  Week 12 | 81.0 (156128.97) | 73.2 (141911.73)
  Week 24 | 73.2 | 71.4

7. Secondary Outcome: Percentage of Participants Who Required Permanent Dose Changes of Study Medication
Time Frame: Week 1 up to Week 24
Population: Per protocol population was a subset of ITT participants who did not have major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 204 | 192
percentage of participants | 86.3 (156128.97) | 93.2 (141911.73)

8. Secondary Outcome: Percentage of Participants Who Required Temporary Dose Changes of Study Medication
Time Frame: Week 1 up to Week 24
Population: Per protocol population was a subset of ITT participants who did not have major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 204 | 192
percentage of participants | 7.4 (156128.97) | 4.2 (141911.73)

9. Secondary Outcome: Percentage of Participants With Any Transient Change of Hemoglobin Level Greater Than (>) 1 Gram Per Deciliter (g/dL)
Time Frame: Week 1 up to Week 24
Population: Per protocol population was a subset of ITT participants who did not have major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 204 | 192
percentage of participants | 44.1 (156128.97) | 43.2 (141911.73)

10. Secondary Outcome: Percentage of Participants With Mean Weekly Hemoglobin Level Outside the Target Range
Description: Percentage of participants who had hemoglobin level outside the target range of 9 to 11 g/dL for the specified weeks were reported.
Time Frame: Week 12, 24
Population: ITT population included all participants who were randomized to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 306 | 306
percentage of participants
  Week 12 | 19.0 | 26.8
  Week 24 | 26.8 | 28.6

11. Secondary Outcome: Percentage of Participants Who Received Blood Transfusions
Time Frame: Week 1 up to Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 303 | 305
percentage of participants | 6.3 (156128.97) | 5.9 (141911.73)

12. Secondary Outcome: Number of Participants With Change in Mean Dose of Study Medication Based on Hemoglobin Level
Description: In this outcome measure number of participants with change (increase and decrease) in mean dose of Epoetin Hospira and Epogen were categorized and reported according to their mean hemoglobin levels. Hemoglobin levels were divided in following classes: >11.0 g/dL, from 9.0 to 11.0 g/dL and <9.0 g/dL
Time Frame: Week 1 up to Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 301 | 305
Participants
  Dose Decrease: Hb <9.0 g/dL | 49 (156128.97) | 37 (141911.73)
  Dose Decrease: Hb (9 to 11 g/dL) | 49 | 46
  Dose Decrease: Hb >11.0 g/dL | 147 | 150
  Dose Increase: Hb <9.0 g/dL | 50 | 67
  Dose Increase: Hb (9 to 11 g/dL) | 27 | 26
  Dose Increase: Hb >11.0 g/dL | 36 | 54

13. Secondary Outcome: Percentage of Participants With Any Transient Change of Hemoglobin Greater Than (>) 2.0 Gram Per Deciliter (g/dL) in Hemoglobin Level
Time Frame: Week 1 up to Week 24
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 301 | 304
percentage of participants | 13.1 (156128.97) | 14.5 (141911.73)

14. Other Pre Specified Outcome: Percentage of Participants With Hemoglobin Level Less Than (<) 8.0 Gram Per Deciliter (g/dL)
Time Frame: Week 1 up to Week 24
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 301 | 304
percentage of participants | 5.3 (156128.97) | 10.9 (141911.73)

15. Other Pre Specified Outcome: Percentage of Participants With Hemoglobin Level Greater Than (>) 12.0 Gram Per Deciliter (g/dL)
Time Frame: Week 1 up to Week 24
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 301 | 304
percentage of participants | 21.6 (156128.97) | 23.0 (141911.73)

16. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; Initial or prolonged in-patient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events from first dose of study drug to the end of study (up to Week 28) that were absent before treatment or that worsened relative to pre-treatment state. AEs included both serious and non-serious adverse events.
Time Frame: Week 1 up to Week 28
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 301 | 304
Participants
  AEs | 232 (156128.97) | 229 (141911.73)
  SAEs | 75 | 82

17. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent were events between first dose of study drug to the end of study (up to Week 28) that were absent before treatment or that worsened relative to pre-treatment state. An AE was assessed according to severity; mild (AE was transient and easily tolerated by the participant), moderate (caused problem that did not interfere significantly with usual activities) and severe (caused problem that interferes significantly with usual activities and might be incapacitating or life-threatening).
Time Frame: Week 1 up to Week 28
Population: Safety population included all participants who received at least 1 dose of study treatment. Here, "N" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 232 | 229
Participants
  Mild | 116 (156128.97) | 111 (141911.73)
  Moderate | 74 | 69
  Severe | 42 | 49

18. Other Pre Specified Outcome: Number of Participants With Treatment Related Adverse Events (AEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug.
Time Frame: Week 1 up to Week 28
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 232 | 229
Participants | 7 (156128.97) | 7 (141911.73)

19. Other Pre Specified Outcome: Number of Participants That Discontinued Treatment Due to a Treatment Emergent Adverse Event
Description: In this outcome measure number of participants who discontinued from study drug (Epoetin Hospira, Epogen) due to any AE were reported.
Time Frame: Week 1 up to Week 28
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 232 | 229
Participants | 9 (156128.97) | 11 (141911.73)

20. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters
Description: Laboratory parameters: Hematology (hematocrit, hemoglobin, red blood cell count, reticulocytes, white blood cell count, neutrophils, bands, lymphocytes, monocytes, basophils, eosinophils, platelet count, mean corpuscular volume); coagulation panel (prothrombin time, international normalized ratio, activated partial thromboplastin time); clinical chemistry (blood urea nitrogen, creatinine, alanine aminotransferase, aspartate aminotransferase, total bilirubin, gamma-glutamyl transpeptidase, alkaline phosphatase, sodium, potassium, calcium, magnesium, phosphorus, uric acid, total protein, glucose, albumin, C-reactive protein, plasma ferritin, transferrin saturation). Participants with clinically significant change from baseline in laboratory parameters were as determined by the investigator.
Time Frame: Baseline up to Week 28
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 301 | 304
Participants | 0 (156128.97) | 0 (141911.73)

21. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital sign parameters: temperature (oral, tympanic, or other), blood pressure (diastolic and systolic), heart rate (in a seated position) and dry weight (post-dialysis). Participants with clinically significant change from baseline in vital signs were as determined by the investigator.
Time Frame: Baseline up to Week 28
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 301 | 304
Participants | 0 (156128.97) | 0 (141911.73)

22. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG)
Description: ECG parameters: PR interval, QRS complex, QT interval and QTC interval. Participants with clinically significant change from baseline in ECG were as determined by the investigator.
Time Frame: Baseline up to Week 28
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 301 | 304
Participants | 0 (156128.97) | 0 (141911.73)

23. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination
Description: Physical examination included examination of the following: skin, eyes, ears, throat, cardiac, respiratory, gastrointestinal, genitourinary and musculoskeletal systems. Participants with clinically significant change from baseline in physical examination were as determined by the investigator.
Time Frame: Baseline up to Week 28
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 301 | 304
Participants | 0 (156128.97) | 0 (141911.73)

24. Other Pre Specified Outcome: Percentage of Participants With Anti-Recombinant Human Erythropoietin (Anti-rhEPO) Antibodies
Description: Percentage of participants with presence of anti-rhEPO antibodies were reported in this outcome measure. Radioimmunoprecipitation assay method was used to determine the presence of anti-rhEPO antibodies.
Time Frame: Week 1 up to Week 28
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 301 | 304
percentage of participants | 0.4 (156128.97) | 0.0 (141911.73)

ADVERSE EVENTS:
Description: Same event may appear as both AE and SAE. What is presented are distinct events. An event may be categorized as serious in 1 participant and as non serious in another participant, or 1 participant may have experienced both a serious and non serious event during the study. Safety population.
Arm/Group | Epoetin Hospira | Epogen
Serious Adverse Events (participants affected / at risk) | 75/301 | 82/304
Other Adverse Events (participants affected / at risk) | 143/301 | 141/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Epoetin Hospira (N=301) | Epogen (N=304)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 2
Angina pectoris (Cardiac disorders) | 1 | 4
Atrial fibrillation (Cardiac disorders) | 2 | 1
Bradycardia (Cardiac disorders) | 3 | 1
Cardiac arrest (Cardiac disorders) | 0 | 3
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 4 | 3
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 2 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 2 | 0
Device malfunction (General disorders) | 1 | 0
Medical device complication (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 7
Pain (General disorders) | 1 | 0
Pelvic mass (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Sudden death (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Arteriovenous graft site infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bursitis infective (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 6
Chest wall abscess (Infections and infestations) | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 2
Device related sepsis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 3
Gastroenteritis (Infections and infestations) | 1 | 1
Graft infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 4 | 8
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 3
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
West Nile viral infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 2
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2 | 2
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/160 | 1/175 — This event was gender specific.
Basal ganglia haemorrhage (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Cervical myelopathy (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 2 | 0
Renal cyst ruptured (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aortic aneurysm (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 2
Hypertensive crisis (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Steal syndrome (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Hospira (N=301) | Epogen (N=304)
Diarrhoea (Gastrointestinal disorders) | 21 | 27
Nausea (Gastrointestinal disorders) | 30 | 25
Vomiting (Gastrointestinal disorders) | 28 | 15
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 25 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 27 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 17
Dizziness (Nervous system disorders) | 19 | 14
Headache (Nervous system disorders) | 23 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 15
Hypertension (Vascular disorders) | 17 | 11
Hypotension (Vascular disorders) | 13 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.